CLINICAL TRIAL: NCT05191758
Title: Nutritional Regulation of Leukocyte Function
Acronym: FPP Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Osato Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Sashwati Roy, Professor of Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13229
Record Dates: First submitted 2021-12-02; First posted 2022-01-13 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: FPP; Fermented Papaya Preparation; Supplements; Diabetic Wound; Healing Wound
Keywords: fermented papaya; wound healing responses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control (No Intervention): no supplements will be taken
- 3 grams of supplements (Experimental): subjects will take 3 grams of supplements once per day
  Interventions: Dietary Supplement: FPP supplement
- 6 grams of supplements (Experimental): subjects will take 3 grams of supplements twice per day
  Interventions: Dietary Supplement: FPP supplement
- 9 grams of supplements (Experimental): subjects will take 3 grams of supplements three times per day
  Interventions: Dietary Supplement: FPP supplement

INTERVENTIONS:
Dietary Supplement: FPP supplement — Participants will take the supplements per randomization
  Other Names: Fermented Papaya Preparation Supplement (FPP); FPP
  Arms: 3 grams of supplements; 6 grams of supplements; 9 grams of supplements

SUMMARY:
The objective of the current study is to determine the dose at which Fermented Papaya Preparation ( FPP) is able to improve inducible respiratory burst outcomes in peripheral blood mononuclear cells (PBMC) and neutrophils of participants. Our investigators have reported that supplementation with standardized fermented papaya preparation (FPP) in mice improves dermal wound healing outcomes. Therefore, based on these observations, the investigators propose to study the dose at which FPP supplementation induces respiratory burst in blood-derived myeloid cells in healthy subjects.

DETAILED DESCRIPTION:
Fermented Papaya Preparation (FPP) is a dietary supplement that is available as over-the-counter in the US. FPP possesses antioxidant properties, which provide benefit against age-related complications[]. Chronic wounds in patients with diabetes represent a major public health problem. Previous studies from the investigators have demonstrated that wound-site macrophages from patients with diabetes are compromised in their ability to support wound healing. Several independent observations convergently point toward the hypothesis that treatment with papaya preparations may facilitate wound healing responses. Our laboratory reported the first evidence demonstrating that FPP may improve diabetic wound outcomes by specifically influencing the response of wound-site macrophages and the subsequent angiogenic response. FPP has a long track record of safe human consumption. The objective of the current study is to determine the dose at which FPP is able to improve inducible respiratory burst outcomes in peripheral blood mononuclear cells (PBMC) and neutrophils of participants. Our investigators have reported that supplementation with standardized fermented papaya preparation (FPP) in mice improves dermal wound healing outcomes. Therefore, based on these observations, the investigators propose to study the dose at which FPP supplementation induces respiratory burst in blood-derived myeloid cells in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and above
* Subjects must be able to follow directions and give informed consent on their own

Exclusion Criteria:

* • Individuals who are deemed unable to understand the procedures, risks and benefits of the study, ie. Informed consent will be excluded.

  * Females who are pregnant will also be excluded to minimize the risk to such individuals (and fetus).
  * Individuals who are therapeutically immuno-compromised will also be excluded to decrease statistical variability and to minimize potential of confounders.
  * Candidates for inclusion into the study will not include individuals as defined in 45 CFR 46 Subparts B, C and D, nor from any other population which may be considered vulnerable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Reactive Oxygen species (ROS) production of Leucocytes 6 weeks post supplementation | 6 weeks post supplementation
  The major objectives of the study is to study the mechanism of action on ROS production by leucocytes of healthy subjects post 6 weeks FPP supplementation measured by flowcytometry
Blood leukocyte phagocytosis 6 weeks post supplementation | 6 weeks post supplementation
  Blood leukocyte phagocytosis 6 weeks post supplementation via cell biology technique

SECONDARY OUTCOMES:
Leukocyte activation and cytokine production at 6 wks post supplementation | 5 weeks
  Blood leukocyte activation and cytokine production at 6 weeks post supplementation will be measured via flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Sashwati Roy, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health Methodist Hospital, Indianapolis, Indiana, United States